CLINICAL TRIAL: NCT05762068
Title: Expert Consensus Statements for the Management of a Physiologically Difficult Airway Using the Delphi Method (PDADelphi)
Acronym: PDADelphi
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kunal Karamchandani, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2023-XXXX
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication; Hemodynamic Instability; Critical Illness
Keywords: Tracheal intubation; Difficult airway; Physiologically Difficult Airway; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Airway management experts: The Steering Committee selected Experts from across the globe based on pre-defined criteria and will conduct iterative Delphi rounds to generate consensus among the experts.
  Interventions: Other: Delphi procedure

INTERVENTIONS:
Other: Delphi procedure — The study involves generating consensus statements by experts on airway management in critically ill patients on the definition and management of a physiologically difficult airway (PDA) using a Delphi process.

SUMMARY:
The aim of this study is to review/identify the existing definition and management strategies for a physiologically difficult airway (PDA), to generate expert consensus on the various aspects of managing a patient with a PDA using the Delphi method, and to provide guidance to clinicians worldwide on safe tracheal intubation practices in patients with PDA to help improve patient outcomes.

DETAILED DESCRIPTION:
The Delphi method involves the following 4 steps:

Step 1: Establishing a preliminary list of broad domains

A focused literature review was performed by select membership of the Society of Critical Care Anesthesiologists (SOCCA), and based on their input, the steering committee identified six broad domains, which were used to draft statements for Round one of the Delphi process.

List of domains:

1. Definitions of PDA
2. Preparing the team for airway management in a patient with PDA
3. Preparing the patient with a PDA for success with airway management
4. Performing tracheal intubation
5. Post-intubation care
6. Areas of Future Research

Step 2: Preparation of the Delphi Round One Survey The list of questions related to the above-mentioned domains will be sent to the Experts as a Delphi questionnaire. The anonymity of the Experts will be maintained during the Delphi rounds. The Experts would be requested to answer questions related to PDA based on their experience and knowledge of the subject. The questions will be multiple choice or in the form of a 7-point Likert scale (strongly agree, agree, somewhat agree, neither agree nor disagree, somewhat disagree, disagree, strongly disagree). The experts can also provide their opinion on addition, deletion on questions or choices through free-text. The responses of experts will be collated during the analysis of results and shared in the following survey as controlled feedback.

Step 3: Subsequent Delphi Rounds The steering committee will review the results of round one. The statements listed will be modified, deleted, or added if found ambiguous based on the feedback and comments of the results. The remaining statements will be continued in the subsequent rounds until consensus is achieved (>80% of respondents). The summary results of round two will be presented to experts, and the survey process will be repeated with the modified questionnaire. The Delphi rounds will be continued till desired consensus and stability is achieved for statements. The steering committee will also check the stability using chi-square test of the statements from Round 3 onwards and statement is said to be stable if p-value is > 0.05 for two consecutive rounds.

Step 4: Final Consensus The summary results of the last stable round will be used to issue the consensus on the various statements related to the above-mentioned domains. The results of the final survey, consensus statements, and the manuscript will be circulated among the experts for approval before submission for publication.

ELIGIBILITY:
Inclusion Criteria:

* Clinical expertise in the airway management of critically ill patients
* Teaching experience in airway management
* Research projects and/or publications in airway management

Exclusion Criteria:

* People don't meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experts must meet the following three criteria:
  Clinical expertise in the airway management of critically ill patients, teaching experience in airway management, and have/had research projects and/or publications in airway management
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Consensus statements | Through study completion, an average of 12 months
  Consensus amongst the expert panel regarding physiologically difficult airway (PDA) management will be achieved using Delphi method which includes iterative rounds of questions.
  Consensus will be considered reached when a statement achieves >80% of votes for multiple-choice questions and >70% for Likert-scale statements.

CONTACTS AND LOCATIONS:
Overall Officials: Kunal Karamchandani, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mosier JM, Joshi R, Hypes C, Pacheco G, Valenzuela T, Sakles JC. The Physiologically Difficult Airway. West J Emerg Med. 2015 Dec;16(7):1109-17. doi: 10.5811/westjem.2015.8.27467. Epub 2015 Dec 8. PMID 26759664
- [Result] Myatra SN, Divatia JV, Brewster DJ. The physiologically difficult airway: an emerging concept. Curr Opin Anaesthesiol. 2022 Apr 1;35(2):115-121. doi: 10.1097/ACO.0000000000001102. PMID 35165233
- [Result] Russotto V, Myatra SN, Laffey JG, Tassistro E, Antolini L, Bauer P, Lascarrou JB, Szuldrzynski K, Camporota L, Pelosi P, Sorbello M, Higgs A, Greif R, Putensen C, Agvald-Ohman C, Chalkias A, Bokums K, Brewster D, Rossi E, Fumagalli R, Pesenti A, Foti G, Bellani G; INTUBE Study Investigators. Intubation Practices and Adverse Peri-intubation Events in Critically Ill Patients From 29 Countries. JAMA. 2021 Mar 23;325(12):1164-1172. doi: 10.1001/jama.2021.1727. PMID 33755076
- [Result] Karamchandani K, Wheelwright J, Yang AL, Westphal ND, Khanna AK, Myatra SN. Emergency Airway Management Outside the Operating Room: Current Evidence and Management Strategies. Anesth Analg. 2021 Sep 1;133(3):648-662. doi: 10.1213/ANE.0000000000005644. PMID 34153007
- [Result] Kornas RL, Owyang CG, Sakles JC, Foley LJ, Mosier JM; Society for Airway Management's Special Projects Committee. Evaluation and Management of the Physiologically Difficult Airway: Consensus Recommendations From Society for Airway Management. Anesth Analg. 2021 Feb 1;132(2):395-405. doi: 10.1213/ANE.0000000000005233. PMID 33060492
- [Result] Diamond IR, Grant RC, Feldman BM, Pencharz PB, Ling SC, Moore AM, Wales PW. Defining consensus: a systematic review recommends methodologic criteria for reporting of Delphi studies. J Clin Epidemiol. 2014 Apr;67(4):401-9. doi: 10.1016/j.jclinepi.2013.12.002. PMID 24581294
- [Result] Nasa P, Jain R, Juneja D. Delphi methodology in healthcare research: How to decide its appropriateness. World J Methodol. 2021 Jul 20;11(4):116-129. doi: 10.5662/wjm.v11.i4.116. eCollection 2021 Jul 20. PMID 34322364